CLINICAL TRIAL: NCT05863533
Title: Resilience,Performance and Stress in Anaesthesia Professionals: a Simulation-based Observational Study
Brief Title: Resilience, Performance and Stress in Anaesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254 - 2023 - 030
Record Dates: First submitted 2023-05-03; First posted 2023-05-18 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Resilience; Stress, Psychological
Keywords: Resilience; Acute stress; Performance; Anaesthetist student; Simulation
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to determine whether there was an association between resilience and the performance of student nurse anaesthetists in simulated critical situations.

DETAILED DESCRIPTION:
This trial will take place at the Grenoble Alpes University Hospital. Volunteer nurse anaesthetists students will perform a simulation scenario. This scenario generates a high level of stress and focuses on the management of anaphylactic shock in the operating room, which is a good teaching tool for the participants.

The simulation is performed in a dedicated simulation room configured as an operating theatre. In this environment, a high-fidelity manikin is intubated and ventilated on an anaesthesia ventilator. The manikin is perfused. The anaesthesia cart is replicated with the same equipment and drugs as the anaesthesia carts in the operating theatre. A person playing the role of a nurse anaesthetist will conduct transmissions before leaving the room replaced by the participant. One person will play the role of the surgeon in the room. The simulation will take place as follows:

Briefing :

Welcome and explanation of the session. Collection of age, gender, number of years in anaesthesia, number of years as a nurse.

The simulation room, the mannequin and the anaesthesia trolley are presented by a simulation trainer before starting the scenario.

First evaluation of the acute stress perceived by the VAS stress(visual analogue stress scale) which triggers the beginning of the scenario.

The patient is introduced by the nurse anaesthetist present in the room and explanations are given on how to reach the anaesthetist by phone. Once the transmissions are completed, the preoperative checklist is carried out by the surgeon with the nurse anaesthetist and the student nurse anaesthetist who takes over. Once the checklist is completed the simulation timer is started and the nurse anaesthetist leaves the room leaving the patient alone on the anaesthesia side.

Scenario:

On arrival at the room:

→ Vitals on arrival: BP (blood pressure)= 100/50, HR(heart rate) = 60, Spo2 = 99%, EtC02 (end tidal C02) = 36 mmHg

T0: Surgical incision

→ Vitals at incision: BP = 120/70, HR = 70, SpO2 = 99%, EtCo2 = 39 mmHg

T1 = 3 min: BP = 90/55, HR = 95, SpO2 = 98%, EtCo2 = 34 mmHg

T2 = 6 min: BP = 78/45, HR = 110, SpO2 = 97%, EtCo2 = 30 mmHg, if possible: vary the SpO2 signal if possible

T3 = 9 min: BP = 65/32, HR = 130, SpO2 = no signal, EtCO2 = 28 mmHg

T4 = 12 min: BP = 56/28, HR = 150, SpO2 = no signal, EtCO2 = 25 mmHg

If no communication with the surgical team before T3, the facilitating surgeon mentions a skin rash to guide management.

The study stops at 12 minutes when the anaesthetist enters the operating room.

Debriefing: The debriefing is conducted by a simulation trainer accordance with the guidelines of the French Society of Health Simulation.

The main objective of this study is to investigate an association between the level of resilience of student nurse anaesthetists and their performance (Performance score N°1) under stress.

The secondary objectives of this study are to investigate the correlation between :

* Performance score N°2 (without taking into account the notion of time in scale N°1) and resilience by ConnorDavison Resilience scale (CDRISC 10).
* Work experience and performance score 1
* Years of specialisation in anesthesia and Performance score 1
* Age and performance score 1

ELIGIBILITY:
Inclusion Criteria:

* Voluntary first or second year nurse anaesthetist student

Exclusion Criteria:

* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurse in the first or second year of specialisation as a nurse anaesthetist.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Resilience | at Day 0 : 10 minutes before simulation
  Measurement of resilience by Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40) in participants. A high score indicates better resilience.

SECONDARY OUTCOMES:
Performance score 1 | at Day 0 during the simulation between T: 0 minute (begin simulation) and T:12 minutes (end of simulation) (during of simulation is 12 minutes))
  Performance scale with 15 items based on the recommendations for the management of anaphylactic shock by the French Society of Anaesthesia and Intensive Care. The time taken to perform the procedure is noted and influences the score. The final score ranges from 0 to 60 points. A higher score indicates a higher performance.
Performance score 2 | at D0 during the simulation between T: 0 minute (begin simulation) and T:12 minutes (end of simulation) (during of simulation is 12 minutes)
  Performance scale with 15 items based on the recommendations for the management of anaphylactic shock by the French Society of Anaesthesia and Intensive Care. The final score ranges from 0 to 15 points. A higher score indicates a higher performance.
Age of anaesthesia professionals | at Day 0 : 10 minutes before simulation
  Age of anesthesia professionals: (quantitative variable)
work experience | at Day 0 : 10 minutes before simulation
  number of years since first nursing practice (quantitative variable)
year of specialisation | at Day 0 : 10 minutes before simulation
  Year of specialisation : first year or second year(qualitative variable)

CONTACTS AND LOCATIONS:
Overall Officials: Julien Picard, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Grenoble Hospital, Grenoble, France